CLINICAL TRIAL: NCT04599374
Title: the Association Between Thyroid Hormones and Metabolic Components in Patients With Obesity
Status: Completed | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Shen Qu, Principal Investigator, Shanghai 10th People's Hospital
Other Study IDs: THs
Record Dates: First submitted 2020-09-29; First posted 2020-10-22 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Obesity; Euthyroid Condition; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- high TSH and high FT4: patients with high TSH and high FT4
  Interventions: Other: no intervention
- high TSH and low FT4: patients with high TSH and low FT4
  Interventions: Other: no intervention
- high TSH and high FT3: patients with high TSH and high FT3
  Interventions: Other: no intervention
- high TSH and low FT3: patients with high TSH and low FT3
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — This study collected data only without any intervention.

SUMMARY:
This study collected clinical data of obese patients with euthyroid function, including age, gender, height, weight, BMI, waist circumference, blood pressure, fasting blood sugar, blood sugar 2 hours after sugar load, fasting plasma high-density lipoprotein cholesterol, fasting three acyl glycerin, free iodine thyroid hormone (FT3) and free thyroid hormones (FT4), thyroid stimulating hormone (TSH), follow-up information and etc. Via analyzing the data, the investigators want to investigate the association between thyroid hormones (THs) and metabolic components in obese patients with euthyroid function and to present the cutoff values of THs in order to provide new information for the risk stratification of metabolic syndrome in obese patients with euthyroid function.

ELIGIBILITY:
Inclusion Criteria:

* 1) age ranged from 18-65 years old, 2) BMI over 27.9kg/m2,3)TSH，FT4, and FT3 within the range of 0.38-4.34mIU/L, 10.5-24.4mIU/L, and 2.8-6.3mIU/L, respectively.

Exclusion Criteria:

* secondary cause of obesity such as hypothalamic obesity, Cushing syndrome, and hypophysis dysfunction, etc.,2)pregnancy or location, 3) severe heart, liver and kidney dysfunction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We enrolled obese patients with euthyroid function.
Sampling Method: Non-Probability Sample
Enrollment: 373 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
meet the criteria of metabolism in the 2017 Chinese guideline | 2015-2020
  1. Abdominal obesity (or central obesity), male abdominal circumference ≥90cm, female abdominal circumference ≥85 cm;
  2. Hypertension, those who have been diagnosed with hypertension and are in treatment and (or) blood pressure ≥130/85mmHg (1mmHg = 0.133kPa);
  3. Hyperglycemia, those who have been diagnosed with diabetes and are treated and (or) fasting blood glucose ≥6.1mmol/L or 2h blood glucose ≥7.8mmol/L after glucose load;
  4. Fasting high-density lipoprotein cholesterol (HDL-C) <1.04mmol/L;
  5. Fasting triacylglycerol ≥1.70mmol/L.

SECONDARY OUTCOMES:
high uric acid | 2015-2020
  female patients with uric acid over 360 umol/L and male female patients with uric acid over 420 umol/L
FBG≥6.1mmol/L | 2015-2020
  patients with fasting blood glucose 6.1mmol/L or more.
BG120≥7.8mmol/L | 2015-2020
  patients with 2 hour blood glucose 7.8mmol/L or more.
FINS≥24.9 pmol/ml | 2015-2020
  patients with fasting insulin 24.9 pmol/ml or more.
FCP≥4.4nmol/L | 2015-2020
  patients with fasting C-peptide 4.4nmol/L or more.

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) are not available to other researchers.